CLINICAL TRIAL: NCT00134498
Title: Phase 3, Multi-Site, Double-Blind, Randomized, Forced Titration, Parallel Group Evaluation Of The Efficacy, Safety, And Tolerability Of Fixed Combination Torcetrapib (CP 529,414)/Atorvastatin Administered Orally, Once Daily (Qd) For Eighteen Weeks, Compared With Atorvastatin Alone, In Subjects With Fredrickson Type IV Hypertriglyceridemia
Brief Title: A Study Comparing The Efficacy & Safety Of Torcetrapib/Atorvastatin And Atorvastatin In Subjects With High Triglycerides
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091025
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-03

CONDITIONS: Hypertriglyceridemia; Hyperlipoproteinemia Type IV
MeSH Terms: conditions — Hypertriglyceridemia; Hyperlipoproteinemia Type IV | interventions — torcetrapib; Atorvastatin

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: atorvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To assess the safety and efficacy of the fixed combination torcetrapib/atorvastatin in subjects with Fredrickson Type IV Hypertriglyceridemia.

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Fredrickson Type IV Hypertriglyceridemia

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects with a clinically indicated need for statin (HMG-CoA reductase inhibitor) therapy other than atorvastatin or other concomitant therapy with known lipid altering effects on LDL-C and HDL-C including fibrates and nicotinic acid
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluation of response, or render unlikely that the subject would complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2005-02; Study Completion 2006-11

PRIMARY OUTCOMES:
Change in HDL-C and non-HDL-C levels

SECONDARY OUTCOMES:
Changes in levels of other lipid and biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (39):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Orangevale, California
  - Pfizer Investigational Site, Pacific Palisades, California
  - Pfizer Investigational Site, Studio City, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Longwood, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Tripler AMC, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Canton, Michigan
  - Pfizer Investigational Site, Portage, Michigan
  - Pfizer Investigational Site, Richland, Michigan
  - Pfizer Investigational Site, Saint Cloud, Minnesota
  - Pfizer Investigational Site, Olive Branch, Mississippi
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, West Seneca, New York
  - Pfizer Investigational Site, Statesville, North Carolina
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Madison, Wisconsin
- Canada (5):
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Ste-Foy, Quebec

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5091025&StudyName=A+Study+Comparing+The+Efficacy+%26+Safety+Of+Torcetrapib%2FAtorvastatin+And+Atorvastatin+In+Subjects+With+High+Triglycerides